CLINICAL TRIAL: NCT01164605
Title: Pilot Study on the Efficacy of a Two Drug, Raltegravir-based Regimen,(NRTI) Sparing Antiretroviral Treatment
Brief Title: Pilot Study of Raltegravir Lipodystrophy IISP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #37977
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infection
Keywords: NRTI-regimen; Raltegravir; Elvitegravir; HIV-1 integrase inhibitor; Fat Waste
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Raltegravir — 60 tablets (30-day supply)

SUMMARY:
The substitution of raltegravir for the NRTIs will result in some reversal of the long term adverse effect of lipodystrophy (specifically peripheral lipoatrophy) that is associated with the chronic use of NRTIs. Changing the HAART regimen in patients with a sustained virological response from a PI plus NRTI to a regimen of the PI plus raltegravir will likely result in continued virologic efficacy.

DETAILED DESCRIPTION:
A prospective, non-controlled, non-randomized, single center study of a treatment regimen of a protease inhibitor or a non-nucleoside reverse transcriptase inhibitor in combination with raltegravir in patients with HIV-1 infection who have been, and continue to be, fully controlled on a standard HAART regimen of a PI or an NNRTI plus 2 NRTIs, and the effect of the change in regimen on peripheral fat distribution.

This pilot study will contain 30 patients who will be followed over a period of one year starting from the date of the medication change from an NRTI-based regimen to a raltegravir-based NRTI-sparing regimen. Potential changes in fat distribution (fat content as assessed by fat volume) will be measured with serial MRI's of the thighs.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 positive
2. Any patient on a boosted PI plus 2 NRTIs.
3. Visual evidence peripheral fat wasting
4. HIV-1 viral load fully suppressed at least 9mths.

Exclusion Criteria:

1. Historical resistance to PI patient receiving
2. No prior exposure to raltegravir, elvitegravir, other HIV-1 integrase inhibitor.
3. No contraindications to serial MRI scanning.
4. No contraindications to utilization of raltegravir.
5. Not currently receiving any medications drug-drug interaction w/ raltegravir.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Determine if the substitution of raltegravir for 2 NRTI's in patients with evidence of peripheral lipoatrophy and who have sustained HIV virological suppression will result in evidence of an increased in volume of peripheral fat within one year. | one year

SECONDARY OUTCOMES:
Determining whether the patients will continue to have sustained virological suppression upon switching to a raltegravir-based regimen. | eighteen months
Determining what, if any, adverse effects the patients may develop.. | eighteen months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Berman, M.D., Ph.D., Principal Investigator — Southern California Institute for Research and Education
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States

REFERENCES:
- [Background] Bickel M, Eisen J, Stephan C, Crespi CM, Lutz T, Klauke S, Vogl TJ, Jacobi V, Yang OO, Staszewski S, Zangos S. A standardized, comprehensive magnetic resonance imaging protocol for rapid and precise quantification of HIV-1-associated lipodystrophy. HIV Med. 2007 Oct;8(7):413-9. doi: 10.1111/j.1468-1293.2007.00487.x. PMID 17760732
- [Background] Efficacy, safety and tolerability of dual therapy with raltegravir and atazanavir in antiretroviral experienced patients. D. Ripamonti, F. Maggiolo, E. Bombana, et al. Presented at the 5th IAS Conference on HIV Pathogenesis, Treatment and Prevention, July 19-22, 2010, Cape Town, South Africa.
- [Background] Raltegravir without a protease inhibitor is highly efficacious in heavily pre-treated individuals. D. Skiest, C. Cohen, D. Barker, M. Gottlieb, et al. Presented at the 5th IAS Conference on HIV Pathogenesis, Treatment and Prevention, July 19-22, 2010, Cape Town, South Africa.
- [Background] Steigbigel RT, Cooper DA, Teppler H, Eron JJ, Gatell JM, Kumar PN, Rockstroh JK, Schechter M, Katlama C, Markowitz M, Yeni P, Loutfy MR, Lazzarin A, Lennox JL, Clotet B, Zhao J, Wan H, Rhodes RR, Strohmaier KM, Barnard RJ, Isaacs RD, Nguyen BY; BENCHMRK Study Teamsa. Long-term efficacy and safety of Raltegravir combined with optimized background therapy in treatment-experienced patients with drug-resistant HIV infection: week 96 results of the BENCHMRK 1 and 2 Phase III trials. Clin Infect Dis. 2010 Feb 15;50(4):605-12. doi: 10.1086/650002. PMID 20085491